CLINICAL TRIAL: NCT03079154
Title: A Pilot RCT Intervention to Test the Impact of High and Low-intensity Mindfulness-based Cognitive Therapy (MBCT) on Self, Values, and Well-being
Brief Title: The Influence of Mindfulness on the Link Between Consumer Culture Values and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sussex (Other)
Collaborators: Sussex Mindfulness Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ER/HELGAD/10
Record Dates: First submitted 2017-03-02; First posted 2017-03-14 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Mental Health and General Well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teacher-led MBCT course (Experimental): Eight-session mindfulness-based cognitive therapy course, including an initial orientation session, led by a qualified mindfulness teacher working with the Sussex Mindfulness Centre, a part of the NHS Sussex Partnership Mental Health Trust.
  Interventions: Other: Teacher-led MBCT course
- Self-guided MBCT course (Active Comparator): Mindfulness-based cognitive therapy course, after an initial information session, which is self-guided using the audiobook Mindfulness: A practical guide to finding peace in a frantic world by Mark Williams and Danny Penman (2011). It consists of eight substantive chapters that map on to the eight-session MBCT course taught by teachers to groups of students. Students will be asked to work through one chapter a week, thus matching the pace of the teacher-led intervention.
  Interventions: Other: Self-guided MBCT course
- Wait list control (No Intervention): Students in the wait list (control) arm do not receive any intervention for the same length of time as the experimental and active comparator arms of the intervention are taking place. Students are invited to complete the self-guided MBCT course after the end of the research project.

INTERVENTIONS:
Other: Teacher-led MBCT course — 9 x 2 hour group sessions following national guidelines for mindfulness-based cognitive therapy
  Other Names: Mindfulness-based cognitive therapy (high intensity)
  Arms: Teacher-led MBCT course
Other: Self-guided MBCT course — 9 weeks of self-guided mindfulness-based cognitive therapy, following an audiobook covering the same material and exercises as the teacher-led intervention
  Other Names: Mindfulness-based cognitive therapy (low intensity)
  Arms: Self-guided MBCT course

SUMMARY:
The study is a three-arm intervention, where students are randomly assigned to one of three conditions: Teacher-led group-based MBCT, Self-guided MBCT using an audio book, or 'wait list' control. Pre-intervention, respondents complete a questionnaire assessing self, values, psychological processes related to self, and well-being. Post-intervention, respondents complete the same questionnaire, and then take part in a laboratory-based study which assesses behaviours related to the variables measured in the questionnaires. We are aiming for a sample size of 180 students at Sussex, 60 in each intervention arm.

DETAILED DESCRIPTION:
Substantive evidence shows that mindfulness training improves mental health and general well-being (see meta-analyses by Cavanagh, Strauss, and colleagues). A significant factor that reduces well-being is the internalisation of two core consumer culture values: a materialistic value orientation (MVO) and body perfect ideals (see meta-analyses by Dittmar and colleagues for MVO, and Grabe et al, Barlett et al. for idealised media models). Thus, mindfulness may act as a buffer against the negative impact of consumer culture ideals, consistent with value circumplex models which place materialistic and appearance-focused values at the self-enhancement end, opposite to self-transcendence values, such as caring for self and others and community engagement.

Self-transcendence values lead to psychological need satisfaction, whereas consumer culture values undermine such satisfaction (Self-Determination Theory).

Three novel questions are examined: (1) Is change in self-related values and psychological processes significant for the beneficial consequences of mindfulness for well-being? (2) Does mindfulness training reduce consumer culture values and associated harmful behaviours, such as disordered eating and excessive buying? (3) Do high and low intensity mindfulness interventions differ in impact?

The project involves collaboration with Kate Cavanagh in Psychology and the Co-Directors of the Sussex Centre for Mindfulness Clara Strauss and Robert Marx. It consists of: 1. qualitative interviews with experienced mindfulness teachers, 2. a multi-phase student intervention study, and 3. an exposure experiment with the same student sample.

Study 1: INTERVIEWS WITH MINDFULNESS TEACHERS (n=12) Semi-structured interviews with teachers (recruited through the UK Network of Mindfulness Teacher Training Organisations) will examine their views on the psychological processes significant in individuals' mental health improvement, focusing on processes related to values and self. Interviews will be audio-taped.

Study 2: INTERVENTION WITH STUDENTS (n=165-180) Phase 1: Online survey to collect baseline measures on all variables of interest, using established scales Trait mindfulness (Gu et al, 2016); Consumer Culture Values (Easterbrook et al., 2014); Core Self Beliefs (Fowler et al, 2006); Self-Discrepancies (Dittmar et al., 1996; Self-compassion (Neff, 2016); Self-esteem (Robins et al., 2001; Self-objectification (Lindner & Tantleff-Dunn, in press); Self-worth (Crocker et al., 2003); Self-concept clarity (Campbell et al., 2003); Self-construal (individualist vs. relational) (Aron et al., 1992); Social comparison tendency (Gibbons & Buunk, 1999); Consumer self-confidence, author, date); Mental health assessment (DASS-21); Subjective well-being (Dittmar & Kapur, 2001); Body esteem (Mendelson et al., 2001); Material esteem (Dittmar et al., 2016); Eating Behaviour (Van Strien et al., 1986, shortened); Excessive Buying (Dittmar et al., 2007); Emotion regulation (Bjureberg, 2016); Consumption-based coping (Wright et al., 2016)

Phase 2: Intervention (randomised control trial)

* 8-week mindfulness-based cognitive group therapy course guided by (non-NHS) mindfulness teachers (high intensity)
* Self-guided MBCT training using a published audio book and CDs (low intensity)
* 'Waiting list' (control; respondents are offered the book after the study)

Phase 3: On-line survey (same as Phase 1) Study 3: IMPACT OF EXPOSURE TO CONSUMER CULTURE STIMULI (n=165-180) Using a 3 (mindfulness intervention condition) x 4 (CC stimuli: materialistic, appearance, combination, control) design, respondents view a film excerpt that contains an ad break (containing CC stimuli, approved in ER/HMC28/2), and then complete measures of actual eating (respondents will be offered food as a reward) and buying behaviour (approved in ER/RLJ/1), as well as selected measures used in Phases 1 and 3.

Studies 2 and 3 include 3 ug and 3 masters research projects.

ELIGIBILITY:
Inclusion Criteria:

Student at the University of Sussex

Exclusion Criteria:

Having experienced a significant life event (e.g., bereavement) in the six months proceeding the study Suffering from a mental health condition at clinical levels Having prior time commitments that prevent the respondents from taking parts in all phases of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Indicators of psychological well-being: Change in Mental health | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  We are using a mental health assessment (DASS-21) widely used in clinical and non-clinical populations which assess symptoms of depression, anxiety, and stress
Indicators of psychological well-being: Change in Subjective well-being | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  This measure consists of an assessment of life satisfaction, and a brief measure of the frequency of positive and negative affective experiences as used in (Dittmar and Kapur, 2011)
Indicators of psychological well-being: Change in consumption-based coping | The change in this self-report measure will be be measured by beingcollected five-six weeks before the intervention, and immediately after the intervention
  This is a newly developed scale which measures the extent to which individuals use buying material goods as a strategy to cope with stress (Wright et. al, 2016)
Indicators of psychological well-being: Change in body esteem | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  We are using a well-established scale of body esteem (Mendelson et al., 2001), which assesses general appearance evaluation, evaluation of one's weight, and perceived evaluation by others
Indicators of psychological well-being: Change in material esteem | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  This is a newly developed scale that assesses individuals' esteem in terms of the material goods they own (Dittmar et al., 2016)
Indicators of psychological well-being: Change in eating behaviour | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  We will use a shortened form of the Dutch Eating Behaviour Scale (Van Strien et al., 1986) which measures restraint, emotional, and external eating
Indicators of psychological well-being: Change in excessive buying | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  This scale measures compulsive buying tendencies, such as having urges to buy or feeling out of control of one's shopping behaviour (Dittmar et al., 2007)
Indicators of psychological well-being: Change in emotional regulation | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  This scale, developed by Bjureberg (2016), assessing difficulties that people experience in dealing with, and regulating strong emotions

SECONDARY OUTCOMES:
Consumer culture values (materialistic and appearance-focused personal values) | This self-report measure will be collected five-six weeks before the intervention, immediately after the intervention, and immediately after exposure to consumer culture stimuli in phase 4 of the research
  This questionnaire measures motives and internalisation with respect to materialistic and appearance-focused values (Easterbrook et al., 2014)
Behavioural measure related to consumer culture: eating | This behavioural measure will be collected immediately after exposure to consumer culture stimuli in phase 4 of the research
  Research participants will be offered a plate of snack foods and told they are can eat as many of them as they would like
Behavioural measure related to consumer culture: buying consumer goods online | This behavioural measure will be collected immediately after exposure to consumer culture stimuli in phase 4 of the research
  Respondents will be invited to use an online retail website for discounted goods to make purchases if they so wish

OTHER OUTCOMES:
Self and self-related processes: Change in core self beliefs | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  Core self beliefs (Fowler et al, 2006) measure the habitual negative and positive beliefs people hold about their self
Self and self-related processes: Change in self-discrepancies | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  Self-discrepancies (Dittmar et al., 1998) refer to perceived gaps between how a person would ideally like to be and how they actually are
Self and self-related processes: Change in self-compassion | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  Self-compassion (Neff, 2016 short form) refers to having a kind and empathic approach to oneself
Self and self-related processes: Change in self-concept clarity | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  Self-concept clarity (Campbell et al., 2003) means that people have a clear and confident view of who and what they are like
Self and self-related processes: Change in self-construal | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  Self-construal (Aron et al., 1992) assesses the extent to which a person sees themselves as an individual entity that is separate for others or connected with others
Self and self-related processes: Change in social comparison tendency | The change in this self-report measure will be be measured by being collected five-six weeks before the intervention, and immediately after the intervention
  Social comparison tendency (Gibbons & Buunk, 1999)

CONTACTS AND LOCATIONS:
Overall Officials: Helga Dittmar, DPhil, Principal Investigator — University of Sussex

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gu J, Strauss C, Crane C, Barnhofer T, Karl A, Cavanagh K, Kuyken W. Examining the factor structure of the 39-item and 15-item versions of the Five Facet Mindfulness Questionnaire before and after mindfulness-based cognitive therapy for people with recurrent depression. Psychol Assess. 2016 Jul;28(7):791-802. doi: 10.1037/pas0000263. Epub 2016 Apr 14. PMID 27078186
- [Background] Easterbrook, M. J., Wright, M. L., Dittmar, H., & Banerjee, R. (2014). Consumer culture ideals, extrinsic motivations, and well-being in children. European Journal of Social Psychology, 44(4), 349-359. doi:10.1002/ejsp.2020
- [Background] Fowler D, Freeman D, Smith B, Kuipers E, Bebbington P, Bashforth H, Coker S, Hodgekins J, Gracie A, Dunn G, Garety P. The Brief Core Schema Scales (BCSS): psychometric properties and associations with paranoia and grandiosity in non-clinical and psychosis samples. Psychol Med. 2006 Jun;36(6):749-59. doi: 10.1017/S0033291706007355. Epub 2006 Mar 27. PMID 16563204
- [Background] Dittmar H, Beattie J, Friese S. Objects, decision considerations and self-image in men's and women's impulse purchases. Acta Psychol (Amst). 1996 Sep;93(1-3):187-206. doi: 10.1016/0001-6918(96)00019-4. PMID 8826795
- [Background] Crocker J, Luhtanen RK, Cooper ML, Bouvrette A. Contingencies of self-worth in college students: theory and measurement. J Pers Soc Psychol. 2003 Nov;85(5):894-908. doi: 10.1037/0022-3514.85.5.894. PMID 14599252
- [Background] Gibbons FX, Buunk BP. Individual differences in social comparison: development of a scale of social comparison orientation. J Pers Soc Psychol. 1999 Jan;76(1):129-42. doi: 10.1037//0022-3514.76.1.129. PMID 9972558
- [Background] Mendelson BK, Mendelson MJ, White DR. Body-esteem scale for adolescents and adults. J Pers Assess. 2001 Feb;76(1):90-106. doi: 10.1207/S15327752JPA7601_6. PMID 11206302
- [Background] Bjureberg J, Ljotsson B, Tull MT, Hedman E, Sahlin H, Lundh LG, Bjarehed J, DiLillo D, Messman-Moore T, Gumpert CH, Gratz KL. Development and Validation of a Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16. J Psychopathol Behav Assess. 2016 Jun;38(2):284-296. doi: 10.1007/s10862-015-9514-x. Epub 2015 Sep 14. PMID 27239096